CLINICAL TRIAL: NCT02216799
Title: Glargine Insulin Versus Continous Regular Insulin in Diabetic Surgical Patients Receiving Parenteral Nutrition (GLUCOSE-in-PN)
Brief Title: Glargine Insulin vs.Continuous Regular Insulin in Diabetic Surgical Patients Receiving Parenteral Nutrition (GLUCOSE-in-PN)
Acronym: GLUCOSE-in-PN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2121166
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Patients With Gastrointestinal Cancer Undergoing Surgery and Receiving Parenteral Nutrition
Keywords: Parenteral nutrition; Hyperglycemia; Glargine insulin; Regular insulin
MeSH Terms: conditions — Hyperphagia; Hyperglycemia; Insulin Resistance | interventions — Insulin Glargine; Injections; Insulin; DNA, Ribosomal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Insulin incorporated in parenteral nutrition (Active Comparator): Regular insulin ( Actrapid, 100 unit/mL0 Solution for injection, Insulin Human (rDNA), Novo Nordisk, will be added to parenteral nutrition to run over 24 hours as 80% of the total insulin requirement of the preceding day administered via subcutaneous sliding scale
  Interventions: Drug: Glargine Insulin; Drug: Regular insulin
- Insulin glargine (Active Comparator): Insulin glargine adminstred at daily night, calculated as 80% of the total insulin requirement of the preceding day from the insulin administered via subcutaneous sliding scale
  Interventions: Drug: Glargine Insulin; Drug: Regular insulin

INTERVENTIONS:
Drug: Glargine Insulin — 80% of the insulin doses administrated via sliding scale will be administered every night as insulin glargine
  Other Names: LANTUS (insulin glargine [rDNA origin] injection
Drug: Regular insulin — 80% of the Regular insulin administrated via sliding scale will be will be added to TPN bag to run over 24 hours
  Other Names: Regular insulin ( Actrapid, 100 unit/mL0 Solution for injection, Insulin Human (rDNA), Novo Nordisk

SUMMARY:
Hyperglycemia increases the risk of complications in surgical patients. Focus on poor glycemic control as a contributor to adverse outcomes in settings outside the intensive care unit (ICU) is often dismissed. Total parenteral Nutrition (TPN) has been used in providing surgical patients with nutrition to prevent deterioration of nutritional status. However, many diabetic patients receiving TPN develop exaggerated hyperglycemia that requires frequent insulin administration via sliding scale. Providing diabetic patient's receiving TPN basal insulin is a known strategy to aid in blood sugar control and prevention of high blood sugar spikes. Many strategies for basal insulin provision have been utilized clinically during the administration of TPN; this includes the incorporation of insulin with TPN solution or administration of long acting insulin such as glargine. However, no study has compared any of these strategies aiming for selecting the optimum modality for controlling blood glucose in diabetic surgical patient's receiving TPN. We will conduct a study to compare the efficacy of once daily insulin glargine versus continuous regular insulin incorporated TPN in controlling blood glucose in non-critically ill diabetic surgical patients receiving TPN.

ELIGIBILITY:
Inclusion Criteria:

* All adult diabetic patients undergoing abdominal surgery operated by the surgical oncology team at KFSH & RC and required TPN therapy are possible subjects of the study.

Exclusion Criteria:

* Patients receiving octreotide or immunosuppressive agents including corticosteroids.
* Recipient of < 3 units of regular insulin per day via subcutaneous insulin sliding scale after the third day of TPN recipient.
* Patients with clinically relevant hepatic disease (> three times normal AST and ALT on admission to the hospital) or impaired renal function (GFR < 60 ml/min), history of diabetic ketoacidosis.

Patients who get infected while on TPN as reflected with elevation of white blood cells and elevated temperature > 37.5 C will be excluded as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Achievement of target blood glucose (140 mg/dL to 200 mg/dL) | 2-years
  Assessemnt of:
  1. Whole blood glucose every morning
  2. The amount of subcutenous insulin adminstraed via sliding scale every 6 hours.
  A target number of 60 patients to complete the study ( 30 patients in each arm) The achievement of target blood glucose based on whole blood glucose levels will be compared in two arms of the study for 5 days while on TPN. Also, the amount of insulin adminstred via sliding scale every day will be comapred as well

SECONDARY OUTCOMES:
Developement of hypoglycemia ( blood glucose < 70 mg/dL) | 2-years
  To assess the development of hypoglycemia in both arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Hakeam A Hakeam, MS., BCPS, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- See also: Study Site — http://www.kfshrc.edu.sa